CLINICAL TRIAL: NCT06893380
Title: A Multicenter Phase 1b/2 Trial Investigating the Efficacy and Toxicity of the Combination of Gemcitabine, Cisplatin, Nab-Paclitaxel, and Tislelizumab in Treatment Naïve Patients With Unresectable, Locally Advanced, or Metastatic BTC
Brief Title: Combination Therapy of GCNT and Tislelizumab in Advanced Biliary Tract Cancer
Acronym: GENTIS
Status: Recruiting | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Hong Jae Chon, Principal Investigator, CHA University
Other Study IDs: CHAMC 2024-09-029
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Biliary Tract Cancers; Metastatic Biliary Tract Cancers
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; 130-nm albumin-bound paclitaxel; tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor tissue and blood samples will be collected and stored for future biomarker analysis, including DNA and RNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combination Therapy Group: This group consists of patients with unresectable, locally advanced, or metastatic biliary tract cancer who will receive combination therapy with Gemcitabine, Cisplatin, Nab-paclitaxel, and Tislelizumab.
  Interventions: Drug: Gemcitabine, Cisplatin, Nab-paclitaxel, and Tislelizumab.

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin, Nab-paclitaxel, and Tislelizumab. — Tislelizumab: IV 200mg on Day 1 of every 3-week cycle Nab-paclitaxel: IV 75mg/m2 on Days 1 and 8 of every 3-week cycle (up to 16 cycles) Gemcitabine: IV 800mg/m2 on Days 1 and 8 of every 3-week cycle Cisplatin: IV 25mg/m2 on Days 1 and 8 of every 3-week cycle (up to 8 cycles)

SUMMARY:
This is a multicenter Phase 1b/2 clinical trial investigating the efficacy and safety of a combination regimen of Gemcitabine, Cisplatin, Nab-paclitaxel, and Tislelizumab in treatment-naïve patients with unresectable, locally advanced, or metastatic biliary tract cancers (BTC), including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer.

The Phase 1b portion aims to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of Nab-paclitaxel in combination with Gemcitabine, Cisplatin, and Tislelizumab. In the Phase 2 portion, the study will evaluate the Objective Response Rate (ORR) as the primary endpoint, with additional assessments of Overall Survival (OS), Progression-Free Survival (PFS), Disease Control Rate (DCR), and Quality of Life (QoL). Safety and tolerability will also be closely monitored.

This study seeks to leverage the stromal-disrupting effect of Nab-paclitaxel and the immune checkpoint blockade effect of Tislelizumab, combined with the established chemotherapy backbone of Gemcitabine and Cisplatin, to enhance treatment outcomes for BTC patients. The study will enroll patients across three medical centers in South Korea, including CHA Bundang Medical Center, Haeundae Paik Hospital, and Seoul National University Bundang Hospital.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) is a heterogeneous group of malignancies arising from the biliary epithelium, including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer. Most patients are diagnosed at unresectable, locally advanced, or metastatic stages, and the prognosis remains poor despite advances in systemic therapy.

Since the ABC-02 trial established Gemcitabine plus Cisplatin as the standard first-line chemotherapy for advanced BTC, numerous combination strategies have been explored to improve survival outcomes. In particular, the addition of Nab-paclitaxel to Gemcitabine and Cisplatin has shown promising efficacy by enhancing stromal penetration and drug delivery, supported by preclinical and early clinical studies.

More recently, immune checkpoint inhibitors (ICIs) have emerged as a new treatment option for BTC. The TOPAZ-1 trial demonstrated that adding Durvalumab to Gemcitabine and Cisplatin significantly improved Overall Survival (OS), establishing immunotherapy-based combination therapy as a new standard of care for advanced BTC. Similarly, the KEYNOTE-966 trial confirmed the benefit of Pembrolizumab combined with Gemcitabine and Cisplatin, further supporting the role of ICIs in BTC management.

Tislelizumab, a humanized PD-1 monoclonal antibody, has shown efficacy in various solid tumors and is now being evaluated in BTC. Compared to other PD-1 inhibitors, Tislelizumab was designed to minimize Fc receptor binding, potentially reducing off-target immune activation and enhancing anti-tumor immune response. Combining Tislelizumab with cytotoxic chemotherapy, including Nab-paclitaxel, may offer synergistic benefits by enhancing antigen release and promoting immune response within the tumor microenvironment.

This Phase 1b/2 multicenter trial aims to investigate the safety, tolerability, and efficacy of the combination regimen of Gemcitabine, Cisplatin, Nab-paclitaxel, and Tislelizumab in treatment-naïve patients with unresectable, locally advanced, or metastatic BTC. The study will be conducted across three medical centers in South Korea: CHA Bundang Medical Center, Haeundae Paik Hospital, and Seoul National University Bundang Hospital.

The Phase 1b part will determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Nab-paclitaxel when combined with Gemcitabine, Cisplatin, and Tislelizumab. Dose escalation will follow a standard 3+3 design, with dose-limiting toxicities (DLTs) assessed during Cycle 1.

In the Phase 2 part, the primary endpoint will be Objective Response Rate (ORR), with secondary endpoints including Overall Survival (OS), Progression-Free Survival (PFS), Disease Control Rate (DCR), Duration of Response (DOR), and Quality of Life (QoL) assessed using EORTC QLQ-C30 and QLQ-BIL21. Safety and tolerability will also be evaluated throughout the study.

This study seeks to optimize the therapeutic potential of chemotherapy plus immunotherapy by incorporating Nab-paclitaxel at a reduced dose to enhance tolerability while maintaining efficacy. Exploratory objectives include assessing immunological and metabolic changes induced by the study drugs, as well as collecting tumor and blood samples for future biomarker analyses.

Through this trial, we aim to establish a novel first-line treatment strategy for advanced BTC, potentially improving survival outcomes beyond the current standard of care.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed biliary tract cancer (BTC), including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer (excluding neuroendocrine tumors, sarcoma, mixed cholangiocarcinoma-HCC, and ampullary carcinoma).
* Age ≥ 19 years at the time of signing informed consent.
* Treatment-naïve for unresectable or metastatic BTC, or recurrence/metastasis at least 6 months after curative surgery or adjuvant chemotherapy.
* Measurable lesions per RECIST v1.1.
* ECOG Performance Status (PS) of 0-1 within 14 days prior to the first dose.
* Life expectancy of ≥ 3 months.
* Adequate organ function (within 14 days prior to the first dose):

  * Hematologic function: Hemoglobin (Hb) ≥ 9.0 g/dL, Absolute neutrophil count (ANC) ≥ 1,500/μL, Platelet count ≥ 100,000/μL
  * Renal function: Serum creatinine ≤ 1.5 × ULN or CrCl (Cockcroft-Gault) ≥ 45 mL/min
  * Hepatic function: AST and ALT ≤ 3.0 × ULN (≤ 5.0 × ULN for hepatic metastases), Total bilirubin ≤ 1.5 × ULN
  * Coagulation: INR ≤ 1.5 or prothrombin time ≤ 1.5 × ULN, aPTT ≤ 1.5 × ULN
* Reproductive status:

  * Female participants must provide proof of non-childbearing status or a negative serum pregnancy test within 7 days before the first dose.
  * Female subjects receiving cisplatin must agree to effective contraception for 14 months after the last dose; male subjects must agree for 11 months.
  * Women of childbearing potential and non-sterilized men must use at least two effective contraceptive methods during the study and for 6 months after the last dose.
* Cardiac function:

  * Left ventricular ejection fraction (LVEF) ≥ 50% (by echocardiography or MUGA scan)
  * No serious valvular disorders or arrhythmias
  * Corrected QT interval ≤ 470 msec at screening
* Willingness to provide tumor tissue samples by biopsy (endoscopic or excisional).

Exclusion Criteria

* Prior treatment history:

  * Prior systemic chemotherapy, biological therapy, immunotherapy, or hormone therapy for unresectable or metastatic BTC
  * Prior adjuvant chemotherapy or radiation therapy within 6 months before recurrence
* History of another malignancy within 5 years, except:

  * Completely resected basal cell carcinoma, stage 1 squamous cell carcinoma, carcinoma in situ, or superficial bladder cancer
* Unresolved toxicities from prior treatment that could affect study evaluation
* Known hypersensitivity to any study drug (tislelizumab, gemcitabine, cisplatin, nab-paclitaxel)
* Active or history of autoimmune disease, except:

  * Hypothyroidism (on stable hormone therapy), vitiligo, or psoriasis not requiring treatment
* History of interstitial lung disease, pulmonary fibrosis, or radiation pneumonitis
* Active gastrointestinal disease:

  * Active peptic ulcer, colitis, or diverticulitis Known central nervous system (CNS) metastasis
* Uncontrolled tumor-related complications: Pericardial effusion, pleural effusion, or ascites requiring intervention, Uncontrolled tumor-related pain
* Significant cardiovascular conditions:

  * Myocardial infarction within 180 days before enrollment
  * Uncontrolled angina within 180 days before enrollment
  * NYHA Class III or IV congestive heart failure
  * Persistent hypertension ≥ 150/90 mmHg despite treatment
  * Arrhythmias requiring medical intervention
  * Thrombosis or vascular diseases requiring surgery
* Uncontrolled diabetes mellitus
* Active infections requiring systemic treatment within 14 days before the first dose
* Recent treatment history:

  * Systemic corticosteroids (except prophylactic or short-term use) or immunosuppressants within 28 days before the first dose
  * Antitumor therapy (cytotoxic, targeted, or immunotherapy) within 28 days before the first dose
  * Pleurodesis within 28 days before the first dose
  * Major surgery under general anesthesia within 28 days before the first dose
  * Local anesthesia or minor surgery within 14 days before the first dose
  * Radiation therapy within 28 days before the first dose (bone metastasis radiation within 14 days is allowed)
* Positive for:

  * HIV-1 or HIV-2
  * Active Hepatitis B or C (except HBV DNA <500 IU/mL with stable antiviral therapy)
* Pregnant or breastfeeding women
* Use of unapproved drugs within 28 days before enrollment
* Cognitive impairment preventing informed consent
* Severe neuropathy (Grade ≥ 2, CTCAE v5.0)
* Hearing impairment
* Inability or unwillingness to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable, locally advanced, or metastatic biliary tract cancer (BTC), including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer, who have not received prior systemic therapy for advanced disease.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months after treatment initiation.
  The proportion of patients who achieve a complete response (CR) or partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 36 months after treatment initiation.
  Time from the date of first dose to the date of death from any cause.
Progression-Free Survival (PFS) | Up to 24 months after treatment initiation.
  Time from the date of first dose to disease progression per RECIST v1.1 or death from any cause.
Disease Control Rate (DCR) | Up to 24 months after treatment initiation.
  The proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) per RECIST v1.1.
Duration of Response (DOR) | Up to 24 months after treatment initiation.
  Time from first documented response (CR or PR) to progression or death.
Quality of Life (QoL)- EORTC QLQ-C30 | Up to 24 months after treatment initiation.
  Patient-reported quality of life assessed using the EORTC QLQ-C30 questionnaire.
Quality of Life (QoL)- EORTC QLQ-BIL21 | Up to 24 months after treatment initiation.
  Patient-reported quality of life assessed using the EORTC QLQ-BIL21 questionnaire.
Safety and Tolerability | Up to 30 days after last dose.
  Incidence, severity, and type of adverse events (AEs), graded per NCI CTCAE v5.0.

OTHER OUTCOMES:
Immune System Response and Immunomodulation Markers | Baseline, during treatment (every 3 cycles; each cycle = 21 days), and at progression (up to 24 months)
  Changes in immune system markers in peripheral blood and tumor tissue samples, including:
  CD8+ T-cell count (%) PD-L1 expression levels in tumor tissues Cytokine levels (e.g., IFN-γ, IL-6, TNF-α) T-cell receptor (TCR) clonality
Metabolic Biomarker Changes in Peripheral Blood and Tumor Tissues | Baseline, during treatment, and at progression (up to 24 months)
  Changes in metabolic biomarkers in peripheral blood and tumor tissue samples, including:
  Serum glucose levels (mg/dL) and insulin resistance markers (e.g., HOMA-IR) Lipid metabolism markers (e.g., triglycerides, total cholesterol, LDL, HDL) Lactate and pyruvate levels as indicators of altered tumor metabolism Amino acid profiling (e.g., glutamine, alanine) for metabolic reprogramming
Collection and Storage of DNA and RNA for Future Exploratory Study | Baseline and during treatment (up to 24 months)
  To collect and store DNA and RNA (following ethical guidelines) for future exploratory research investigating genetic variations that may affect responses to study treatment (distribution, safety, tolerability, and efficacy) and/or susceptibility to diseases. Participation in this exploratory study is optional.
Quality of Life (QoL) - EORTC QLQ-C30 | Baseline, every 3 cycles during treatment (each cycle = 21 days), and at the end of treatment (up to 24 months)
  Patient-reported quality of life assessed using the EORTC QLQ-C30 questionnaire, which evaluates physical, emotional, cognitive, and social functioning.
Quality of Life (QoL) - EORTC QLQ-BIL21 | Baseline, every 3 cycles during treatment (each cycle = 21 days), and at the end of treatment (up to 24 months)
  Patient-reported quality of life specific to biliary tract cancer, assessed using the EORTC QLQ-BIL21 questionnaire, which measures biliary cancer-related symptoms such as jaundice, pain, and fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, MD. PhD, Principal Investigator — Principal Investigator
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sirica AE, Gores GJ. Desmoplastic stroma and cholangiocarcinoma: clinical implications and therapeutic targeting. Hepatology. 2014 Jun;59(6):2397-402. doi: 10.1002/hep.26762. Epub 2014 Apr 9. No abstract available. PMID 24123296
- [Background] Coulouarn C, Clement B. Stellate cells and the development of liver cancer: therapeutic potential of targeting the stroma. J Hepatol. 2014 Jun;60(6):1306-9. doi: 10.1016/j.jhep.2014.02.003. Epub 2014 Feb 12. PMID 24530649
- [Background] Claperon A, Mergey M, Aoudjehane L, Ho-Bouldoires TH, Wendum D, Prignon A, Merabtene F, Firrincieli D, Desbois-Mouthon C, Scatton O, Conti F, Housset C, Fouassier L. Hepatic myofibroblasts promote the progression of human cholangiocarcinoma through activation of epidermal growth factor receptor. Hepatology. 2013 Dec;58(6):2001-11. doi: 10.1002/hep.26585. Epub 2013 Oct 25. PMID 23787814
- [Background] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Background] Oh DY, Ruth He A, Qin S, Chen LT, Okusaka T, Vogel A, Kim JW, Suksombooncharoen T, Ah Lee M, Kitano M, Burris H, Bouattour M, Tanasanvimon S, McNamara MG, Zaucha R, Avallone A, Tan B, Cundom J, Lee CK, Takahashi H, Ikeda M, Chen JS, Wang J, Makowsky M, Rokutanda N, He P, Kurland JF, Cohen G, Valle JW. Durvalumab plus Gemcitabine and Cisplatin in Advanced Biliary Tract Cancer. NEJM Evid. 2022 Aug;1(8):EVIDoa2200015. doi: 10.1056/EVIDoa2200015. Epub 2022 Jun 1. PMID 38319896
- [Background] Piha-Paul SA, Oh DY, Ueno M, Malka D, Chung HC, Nagrial A, Kelley RK, Ros W, Italiano A, Nakagawa K, Rugo HS, de Braud F, Varga AI, Hansen A, Wang H, Krishnan S, Norwood KG, Doi T. Efficacy and safety of pembrolizumab for the treatment of advanced biliary cancer: Results from the KEYNOTE-158 and KEYNOTE-028 studies. Int J Cancer. 2020 Oct 15;147(8):2190-2198. doi: 10.1002/ijc.33013. Epub 2020 May 2. PMID 32359091
- [Background] Kim RD, Chung V, Alese OB, El-Rayes BF, Li D, Al-Toubah TE, Schell MJ, Zhou JM, Mahipal A, Kim BH, Kim DW. A Phase 2 Multi-institutional Study of Nivolumab for Patients With Advanced Refractory Biliary Tract Cancer. JAMA Oncol. 2020 Jun 1;6(6):888-894. doi: 10.1001/jamaoncol.2020.0930. PMID 32352498
- [Background] Shroff RT, King G, Colby S, Scott AJ, Borad MJ, Goff L, Matin K, Mahipal A, Kalyan A, Javle MM, El Dika I, Tan B, Cheema P, Patel A, Iyer R, Kelley RK, Thumar J, El-Khoueiry A, Guthrie KA, Chiorean EG, Hochster H, Philip PA. SWOG S1815: A Phase III Randomized Trial of Gemcitabine, Cisplatin, and Nab-Paclitaxel Versus Gemcitabine and Cisplatin in Newly Diagnosed, Advanced Biliary Tract Cancers. J Clin Oncol. 2025 Feb 10;43(5):536-544. doi: 10.1200/JCO-24-01383. Epub 2024 Dec 13. PMID 39671534
- [Background] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404